CLINICAL TRIAL: NCT02914925
Title: The Effect of Combined Armeospring Pediatric and Constraint Induced Therapy on Neuro-motor and Functional Recovery in Children With Unilateral Cerebral Palsy
Brief Title: The Effect of Combined Armeospring and CIT on Neuro-motor and Functional Recovery in Children With Unilateral CP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Mary's Hospital for Children (Other)
Responsible Party: Principal Investigator, William Watson, Neuropsychologist, St Mary's Hospital for Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMH-001
Record Dates: First submitted 2016-09-21; First posted 2016-09-26 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Cerebral Palsy; Hemiplegia; Upper Extremity Weakness
Keywords: CIT; ArmeoSpring; TMS
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ArmeoSpring/CIT (Experimental): Group will receive ArmeoSpring and CIT therapy
  Interventions: Device: ArmeoSpring/CIT

INTERVENTIONS:
Device: ArmeoSpring/CIT — Participating group will receive therapy with the Armeo®Spring Pediatric and CIT for 6 hours per day, 5 days per week for three weeks, totaling 90 hours

SUMMARY:
The purpose of this study is to assess the use of a commercially available arm weight supporting training system (Armeo®Spring) in conjunction with Constraint Induced Therapy (CIT) for improving upper extremity function for children with unilateral cerebral palsy. In addition, the study aims to assess the potential cortical changes with Armeo®Spring therapy and CIT with the use of the Transcranial Magnetic Stimulation (TMS) motor mapping.

This within-subjects repeated-measures study will be conducted at St. Mary's Hospital for Children. Subjects will be recruited from the general population. A sample size of 10 participants is required for the study. Minority and gender distributions of this study are expected to reflect the distributions in the general population of this region.

Therapy: Participating children will have their unaffected arm placed in a sling. The sling is placed at the start of the day and the child is encouraged to have this on during all therapy sessions.The affected arm will be used for repetitive therapeutic activities.Therapy sessions will include activities aimed at building motor learning skills.

TMS will be used to map the brain. Participants will have MRI of the brain that is T1 weighted with 0.9 -1.1 voxel. size to allow for on-screen navigation of the cerebral cortex while performing TMS.The stimulating coil will be held to the scalp over each M1 hemisphere and an induced electrical current passed through the coil will create a magnetic pulse that stimulates the brain

Children will be assessed using functional hand tests and TMS.

DETAILED DESCRIPTION:
Objective: This study will evaluate the effect of combined Armeo®spring pediatric and Constraint Induced Therapy on neuro-motor and functional recovery in children with unilateral cerebral palsy.

Background: Children with unilateral cerebral palsy (CP) tend not to use their impaired arm and hand throughout life. This disuse of a limb during postnatal development can stunt the activity-dependent structural and functional development of the motor system. Enabling young children to more readily use their affected extremity is likely to increase the competitive ability of the affected side and can improve the functional and anatomical integrity of the motor system.

Several studies have shown that applying a restraint to the less affected hand with intensive repetitive use of the more affected hand has significant effect in overcoming learned non-use. There is evidence that suggests that CIT produced significant cortical reorganization in adults with chronic and sub-acute cerebrovascular accident (CVA) and patients with chronic traumatic brain injury and for the lower limb of patients with CVA.

The associations between motor physiology and motor performance in children with hemiplegic CP are being examined. Recent study shows that children whose impaired hand is controlled by contralateral connections from the unaffected motor cortex show greater improvement to intensive hand training than children whose impaired hand is controlled by ipsilateral connections from the affected motor cortex.

In order for future therapies to be applied selectively to brain regions most important in mediating recovery, it is important to determine the location of plastic changes produced by intensive practice.

Subject Population: Children with CP Hemiplegia

Design: Participating children enrolled will engage in intensive CI therapeutic activities along with 30-45 minutes of Armeo®Spring based activities at progressively increasing levels of difficult, 6 h/day for 5 days a week for three weeks. Each child's performance will be tracked and activities will be modified based on performance.

Hand function would be assessed using functional hands test (AHA, Box & Blocks test, Jebsen Taylor hand function test) and TMS at three time points: before, after and six months after completion of the training protocol.

Outcome measures: Outcome variables of TMS will be measures of corticomotor excitability using single-pulse TMS. Motor evoked potentials (MEPs) will be recorded via surface electromyography (EMG).

Significance: Understanding how rehabilitation can modulate brain areas associated with motor deficits in CP.

ELIGIBILITY:
Inclusion Criteria:

* Children with diagnosis of CP hemiplegia
* Children that meet Armeo®Spring Pediatric fit criteria
* Upper arm measures:155mm-235mm (7 to 9.5 inches)
* Lower arm measures: 230mm-370mm
* Children that have the ability to follow instructions.

Exclusion Criteria:

* Severe cognitive deficits
* Children with any current medical illness unrelated to CP
* Children with previous episode of neurocardiogenic syncope
* Children with visual problems uncorrected by glasses and contact lens
* History of Botulinum toxin or surgical intervention to the relevant extremity in the previous 6 months
* Children with severe spasticity
* Children with severe spontaneous movements-ataxia, myoclonic jerks, dyskinesia
* History of seizure beyond age 2
* History of bone instability, shoulder joint subluxation or pain
* Any child on anti-seizure medications or history of epilepsy in self or first degree relatives
* Any child who has serious heart disease, structural brain lesion,increased intracranial pressure, or has had brain surgery Any child with metals in the body such as cranial metal implants, pacemaker, medication pump, cochlear implant, implanted brain stimulator

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change in motor cortical map expansion | Baseline (within week prior to 3-week intervention), Post-intervention (up to 1 week after 3 week therapy intervention is completed) and 6 months after therapy
  Transcranial Magnetic Stimulation (TMS)
Change in hand function | Baseline (within week prior to 3-week intervention), Post-intervention (up to 1 week after 3 week therapy intervention is completed) and 6 months after therapy
  Box and Blocks test
Change in hand function | Baseline (within week prior to 3-week intervention), Post-intervention (up to 1 week after 3 week therapy intervention is completed) and 6 months after therapy
  Jebsen Taylor Hand Function Test
Change in bimanual hand function | Baseline (within week prior to 3-week intervention), Post-intervention (up to 1 week after 3 week therapy intervention is completed) and 6 months after therapy
  Assisting Hand Assessment

CONTACTS AND LOCATIONS:
Overall Officials: William Watson, Ph.D, Principal Investigator — St Mary's Hospital for Children; Swetha Krishnaswamy, MS OTR/L, Principal Investigator — St Mary's Hospital for Children
Locations (1):
- William Watson, Queens, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Liepert J, Bauder H, Wolfgang HR, Miltner WH, Taub E, Weiller C. Treatment-induced cortical reorganization after stroke in humans. Stroke. 2000 Jun;31(6):1210-6. doi: 10.1161/01.str.31.6.1210. PMID 10835434
- [Background] Inguaggiato E, Sgandurra G, Perazza S, Guzzetta A, Cioni G. Brain reorganization following intervention in children with congenital hemiplegia: a systematic review. Neural Plast. 2013;2013:356275. doi: 10.1155/2013/356275. Epub 2013 Dec 3. PMID 24367726